CLINICAL TRIAL: NCT01990768
Title: Prehospital Tranexamic Acid Use for Traumatic Brain Injury
Acronym: TXA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); U.S. Army Medical Research and Development Command (U.S. Federal Agency); Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other); American Heart Association (Other); Defence Research and Development Canada (Industry)
Responsible Party: Principal Investigator, Susanne May, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 47114; 5U01HL077863-09 (NIH); TATRC Log No. 13335004-A (Other Grant/Funding Number: US Army Medical Research Acquisition Activity (USAMRAA))
Record Dates: First submitted 2013-10-30; First posted 2013-11-21 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-12

CONDITIONS: Traumatic Brain Injury
Keywords: tranexamic acid; traumatic brain injury; intracranial hemorrhage; prehospital; neurologic outcome; glasgow outcome scale extended; disability rating scale
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hemorrhages | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 gram Tranexamic Acid (TXA) (Experimental): Loading dose of 1 gram TXA given prior to hospital arrival followed by a 1 gram TXA infusion over 8 hours after hospital arrival
  Interventions: Drug: 1 gram Tranexamic Acid (TXA)
- 2 grams TXA (Experimental): Loading dose of 2 gram TXA given prior to hospital arrival followed by a placebo of 0.9% Sodium Chloride solution infusion over 8 hours after hospital arrival
  Interventions: Drug: 2 grams TXA
- 0.9% Sodium Chloride injectable (Placebo Comparator): Loading dose of 0.9% Sodium Chloride solution given prior to hospital arrival followed by a placebo of 0.9% Sodium Chloride solution infusion over 8 hours after hospital arrival
  Interventions: Drug: 0.9% Sodium Chloride injectable

INTERVENTIONS:
Drug: 1 gram Tranexamic Acid (TXA) — TXA produces an antifibrinolytic effect by competitively inhibiting the activation of plasminogen to plasmin.
  Other Names: Cyklokapron
  Arms: 1 gram Tranexamic Acid (TXA)
Drug: 2 grams TXA — TXA produces an antifibrinolytic effect by competitively inhibiting the activation of plasminogen to plasmin.
  Other Names: Cyklokapron
  Arms: 2 grams TXA
Drug: 0.9% Sodium Chloride injectable — Loading dose of 0.9% Sodium Chloride solution given prior to hospital arrival followed by a placebo of 0.9% Sodium Chloride solution infusion over 8 hours after hospital arrival. No active drug is added to the solution.
  Other Names: Normal saline solution
  Arms: 0.9% Sodium Chloride injectable

SUMMARY:
Primary aim: To determine the efficacy of two dosing regimens of TXA initiated in the prehospital setting in patients with moderate to severe TBI (GCS score ≤12).

Primary hypothesis: The null hypothesis is that random assignment to prehospital administration of TXA in patients with moderate to severe TBI will not change the proportion of patients with a favorable long-term neurologic outcome compared to random assignment to placebo, based on the GOS-E at 6 months.

Secondary aims: To determine differences between TXA and placebo in the following outcomes for patients with moderate to severe TBI treated in the prehospital setting with 2 dosing regimens of TXA:

* Clinical outcomes: ICH progression, Marshall and Rotterdam CT classification scores, DRS at discharge and 6 months, GOS-E at discharge, 28-day survival, frequency of neurosurgical interventions, and ventilator-free, ICU-free, and hospital-free days.
* Safety outcomes: Development of seizures, cerebral ischemic events, myocardial infarction, deep venous thrombosis, and pulmonary thromboembolism.
* Mechanistic outcomes: Alterations in fibrinolysis based on fibrinolytic pathway mediators and degree of clot lysis based on TEG.

Inclusion: Blunt and penetrating traumatic mechanism consistent with TBI with prehospital GCS ≤ 12 prior to administration of sedative and/or paralytic agents, prehospital SBP ≥ 90 mmHg, prehospital intravenous (IV) access, age ≥ 15yrs (or weight ≥ 50kg if age is unknown), EMS transport destination based on standard local practices determined to be a participating trauma center.

Exclusion: Prehospital GCS=3 with no reactive pupil, estimated time from injury to start of study drug bolus dose >2 hours, unknown time of injury, clinical suspicion by EMS of seizure activity, acute MI or stroke or known history, to the extent possible, of seizures, thromboembolic disorders or renal dialysis, CPR by EMS prior to randomization, burns > 20% TBSA, suspected or known prisoners, suspected or known pregnancy, prehospital TXA or other pro-coagulant drug given prior to randomization, subjects who have activated the "opt-out" process when required by the local regulatory board.

A multi-center double-blind randomized controlled trial with 3 treatment arms:

* Bolus/maintenance: 1 gram IV TXA bolus in the prehospital setting followed by a 1 gram IV maintenance infusion initiated on hospital arrival and infused over 8 hours.
* Bolus only: 2 grams IV TXA bolus in the prehospital setting followed by a placebo maintenance infusion initiated on hospital arrival and infused over 8 hours.
* Placebo: Placebo IV bolus in the prehospital setting followed by a placebo maintenance infusion initiated on hospital arrival and infused over 8 hours.

DETAILED DESCRIPTION:
1. Overview This multi-center, Phase II trial is designed to determine if Tranexamic Acid (TXA) initiated in the prehospital setting improves long-term neurologic outcome compared to placebo in patients with moderate to severe TBI who are not in shock. This study protocol will be conducted as part of the Resuscitation Outcomes Consortium (ROC) at trauma centers in the United States and Canada. ROC is funded by the National Heart Lung and Blood Institute (NHLBI) in partnership with the US Army Medical Research and Materiel Command (USAMRMC), Canadian Institutes of Health Research, the Heart & Stroke Foundation of Canada, the American Heart Association (AHA), and the Defense Research and Development Canada. ROC is a clinical trials network focusing on research primarily in the area of prehospital cardiopulmonary arrest and severe traumatic injury. The mission of ROC is to provide infrastructure and project support for clinical trials and other outcome-oriented research in the areas of cardiopulmonary arrest and severe traumatic injury that lead to evidence-based change in clinical practice.
2. Specific Aims/Hypothesis Statement

   2.1 Clinical Hypotheses and Aims

   Specific aim 1: To compare 6-month neurologic outcome between subjects who are randomly assigned to TXA to subjects who are randomly assigned to placebo by evaluating the Glasgow Outcome Scale Extended score (GOS-E) at 6 months post-injury.

   Primary Hypotheses: We will perform a one-sided test of the following null hypothesis: The proportion of subjects who have a favorable neurologic outcome (GOS-E > 4) at six months post injury who are randomly assigned to TXA is not different from the proportion of subjects who have a favorable neurologic outcome (GOS-E > 4) who are randomly assigned to placebo. This hypothesis will be tested versus the alternative that the proportion of subjects with a favorable neurologic outcome who are randomly assigned to TXA is higher than in subjects who are randomly assigned to placebo at the .1 level and versus the alternative that the proportion of subjects with a favorable neurologic outcome who are randomly assigned to TXA is lower than it is in the placebo group at the .025 level

   Specific aim 2: To assess differences in morbidity and mortality measured from randomization through 28 days or initial hospital discharge and differences in neurologic outcomes at 6 months between subjects in the bolus/maintenance arm, bolus only arm, and placebo arm.

   Secondary Hypotheses: The null hypotheses are that there will be no difference between subjects who are randomly assigned to TXA and subjects who are randomly assigned to placebo in the following: both absolute and relative volume of intracranial hemorrhage (ICH) progression, proportion of subjects with ICH progression, frequency of neurosurgical interventions, GOS-E measured at discharge and 6 months, Disability Rating Scale score (DRS) measured at discharge and 6 months, 28-day survival, and ventilator-free, intensive care unit (ICU)-free, and hospital-free days.

   Specific aim 3: To assess differences in adverse events measured from randomization to initial hospital discharge between subjects in the bolus/maintenance arm, bolus only arm, and placebo arm.

   Tertiary Hypotheses: The null hypotheses are that there will be no difference between subjects who are randomly assigned to TXA and subjects who are randomly assigned to placebo in the following: proportion of subjects experiencing seizures, cerebral ischemic events, myocardial infarction (MI), deep venous thrombosis (DVT), or pulmonary thromboembolism (PE) post randomization through 28 days or discharge, whichever occurs first.

   2.2 Laboratory Hypotheses and Aims

   Specific aim 1: To compare coagulation profiles over time using kaolin activated thrombelastography (TEG) results between subjects who are randomly assigned to TXA and subjects who are randomly assigned to placebo.

   Primary hypothesis: The null hypothesis is that there will be no difference in the degree of fibrinolysis as assessed by percentage of clot lysis determined 30 minutes after the maximum amplitude is reached (LY30) between subjects who are randomly assigned to TXA and subjects who are randomly assigned to placebo.

   Specific aim 2: To explore the underlying mechanism of TXA by comparing fibrinolytic pathway mediator activity between subjects who are randomly assigned to TXA and subjects who are randomly assigned to placebo.

   Secondary hypothesis: The null hypothesis is that there will be no change in fibrinolytic pathway mediators between subjects who are randomly assigned to TXA and subjects who are randomly assigned to placebo.

   Specific aim 3: To estimate the association between the degree of fibrinolysis based on kaolin activated TEG results and fibrinolytic pathway mediators on primary and secondary clinical outcomes.

   Tertiary hypothesis: The null hypothesis is that no association will exist between the degree of fibrinolysis and fibrinolytic pathway mediators and primary and secondary clinical outcomes.
3. Study Enrollment

   EMS agencies will carry blinded sealed study drug kits. Once the seal is broken in the presence of the patient, the patient is randomized. The EMS study drug kit will contain a vial of either 1 gram TXA, 2 grams TXA, or placebo. EMS will mix the study drug in a 250 mL bag of 0.9% sodium chloride and administer the bolus infusion as soon as life-saving interventions are performed. After randomization, EMS will provide the study drug kit ID# to the receiving pharmacy. The hospital pharmacist will obtain the randomization assignment from the coordinating center and prepare the appropriate drug to be administered in the hospital.
4. Sample Size and Statistical Analysis

   The total sample size is 963 (321 per group) starting treatment, which will allow for 80% power to detect a 7.1% absolute difference in favorable long-term neurological outcome as determined by the GOS-E 6 months after injury comparing the combined TXA treatment groups to placebo, using a one-sided, level 0.1 test.

   Statistical analysis of primary hypothesis: Modified intention-to-treat analysis using logistic regression to test for association and estimate the strength of the association of treatment group with a favorable 6-month outcome (defined as a GOS-E > 4), after adjustment for study site.
5. Human subjects protection

This study qualifies for the exception from informed consent (EFIC) required for emergency research outlined in FDA regulation 21CFR50.24. EFIC applies because of life-threatening situation, intervention must be administered before consent is feasible, no reasonable way to identify prospectively individuals at risk, patients have the prospect of benefit from the treatment, and the research could not practically be carried out without the waiver of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Blunt or penetrating traumatic mechanism consistent with traumatic brain injury
2. Prehospital Glasgow Coma Score (GCS) score ≤ 12 at any time prior to randomization and administration of sedative and/or paralytic agents
3. Prehospital systolic blood pressure (SBP) ≥ 90 mmHg prior to randomization
4. Prehospital intravenous (IV) or intraosseous (IO) access
5. Estimated Age ≥ 15 (or estimated weight > 50 kg if age is unknown)
6. Emergency Medicine System (EMS) transport to a participating trauma center

Exclusion Criteria:

1. Prehospital GCS=3 with no reactive pupil
2. Estimated time from injury to hospital arrival > 2 hours
3. Unknown time of injury - no known reference times to support estimation
4. Clinical suspicion by EMS of seizure activity or known history of seizures, acute myocardial infarction (MI) or stroke
5. Cardio-pulmonary resuscitation (CPR) by EMS prior to randomization
6. Burns > 20% total body surface area (TBSA)
7. Suspected or known prisoners
8. Suspected or known pregnancy
9. Prehospital TXA given prior to randomization
10. Subjects who have activated the "opt-out" process when required by the local regulatory board

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 967 (Actual)
Dates: Start 2015-05; Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne May, PhD, Principal Investigator — University of Washington; Martin Schreiber, MD FACS, Principal Investigator — Oregon Health and Science University
Locations (12):
- United States (10):
  - Alabama Resuscitation Center, Birmingham, Alabama
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - St Paul Regions Hospital, Saint Paul, Minnesota
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - Dallas Center for Resuscitation Research, Dallas, Texas
  - Memorial Hermann Hospital - Texas Medical Center, Houston, Texas
  - Harborview Medical Center, Seattle, Washington
  - Milwaukee Resuscitation Research Center, Milwaukee, Wisconsin
- Canada (2):
  - British Columbia Regional Coordinating Center, Vancouver, British Columbia
  - Toronto RescuNet, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Public use data set will be shared with NHLBI. It will include individual patient data that are de-identified. It will be available 3 years after study completion. This is currently expected for the end of 2020. The data should then be available at <https://biolincc.nhlbi.nih.gov/studies/>.

REFERENCES:
- [Derived] Rowell S, Meier EN, Hoyos Gomez T, Fleming M, Jui J, Morrison L, Bulger E, Sopko G, Weisfeldt M, Christenson J, Klotz P, McMullan J, Callum J, Sheehan K, Tibbs B, Aufderheide T, Cotton B, Gandhi R, Idris A, Frascone RJ, Ferrara M, Richmond N, Kannas D, Schlamp R, Robinson B, Dries D, Tallon J, Hendrickson A, Gamber M, Garrett J, Simonson R, McKinley WI, Schreiber M. The effects of prehospital TXA on mortality and neurologic outcomes in patients with traumatic intracranial hemorrhage: A subgroup analysis from the prehospital TXA for TBI trial. J Trauma Acute Care Surg. 2024 Oct 1;97(4):572-580. doi: 10.1097/TA.0000000000004354. Epub 2024 Apr 30. PMID 38685481
- [Derived] Hoefer LE, Benjamin AJ, Polcari AM, Schreiber MA, Zakrison TL, Rowell SE. TXA does not affect levels of TBI-related biomarkers in blunt TBI with ICH: A secondary analysis of the prehospital TXA for TBI trial. J Trauma Acute Care Surg. 2024 Jan 1;96(1):94-100. doi: 10.1097/TA.0000000000004130. Epub 2023 Oct 9. PMID 37807179
- [Derived] Harmer JW, Dewey EN, Meier EN, Rowell SE, Schreiber MA. Tranexamic acid is not inferior to placebo with respect to adverse events in suspected traumatic brain injury patients not in shock with a normal head computed tomography scan: A retrospective study of a randomized trial. J Trauma Acute Care Surg. 2022 Jul 1;93(1):98-105. doi: 10.1097/TA.0000000000003635. Epub 2022 Mar 28. PMID 35358154
- [Derived] Rowell SE, Meier EN, McKnight B, Kannas D, May S, Sheehan K, Bulger EM, Idris AH, Christenson J, Morrison LJ, Frascone RJ, Bosarge PL, Colella MR, Johannigman J, Cotton BA, Callum J, McMullan J, Dries DJ, Tibbs B, Richmond NJ, Weisfeldt ML, Tallon JM, Garrett JS, Zielinski MD, Aufderheide TP, Gandhi RR, Schlamp R, Robinson BRH, Jui J, Klein L, Rizoli S, Gamber M, Fleming M, Hwang J, Vincent LE, Williams C, Hendrickson A, Simonson R, Klotz P, Sopko G, Witham W, Ferrara M, Schreiber MA. Effect of Out-of-Hospital Tranexamic Acid vs Placebo on 6-Month Functional Neurologic Outcomes in Patients With Moderate or Severe Traumatic Brain Injury. JAMA. 2020 Sep 8;324(10):961-974. doi: 10.1001/jama.2020.8958. PMID 32897344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2015 and March 2017, participants were enrolled by 39 emergency management service (EMS) agencies and transported to 20 trauma centers within 12 regional sites in North America.
Pre-assignment Details: Some persons for whom the blinded study kit was opened did not actually receive any of the study drug. These persons are not included in the enrollment numbers. However, they are enumerated in the first section of the patient flow tables.
Groups:
- Placebo: Placebo IV bolus in the prehospital setting followed by a placebo maintenance infusion initiated on hospital arrival and infused over 8 hours.
- Bolus-Maintenance: 1 gram IV TXA bolus in the prehospital setting followed by a 1 gram IV maintenance infusion initiated on hospital arrival and infused over 8 hours.
- Bolus Only: 2 grams IV TXA bolus in the prehospital setting followed by a placebo maintenance infusion initiated on hospital arrival and infused over 8 hours.
Period: Intervention Started
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Started | 345 | 345 | 373
Completed | 309 | 312 | 346
Not Completed | 36 | 33 | 27
Not completed — Found to be ineligible | 14 | 13 | 11
Not completed — Study drug issue or kit malfunction | 9 | 6 | 7
Not completed — Patient became ineligible due to vitals | 5 | 5 | 2
Not completed — Not enough time for EMS to enroll | 4 | 3 | 0
Not completed — Patient care priority | 1 | 2 | 3
Not completed — IV lost | 2 | 2 | 2
Not completed — Required CPR | 1 | 1 | 0
Not completed — Seizure or hx of seizure | 0 | 0 | 2
Not completed — Discovered to be pregnant | 0 | 1 | 0
Period: Prehospital Study Drug Infusion
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Started | 309 | 312 | 346
Completed | 290 | 285 | 327
Not Completed | 19 | 27 | 19
Not completed — Protocol non-compliance | 4 | 11 | 10
Not completed — Seizure or concern for seizure | 4 | 3 | 4
Not completed — Required CPR | 2 | 6 | 0
Not completed — Other safety concern | 2 | 1 | 1
Not completed — Death | 3 | 1 | 1
Not completed — Discharged | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Emergency unblinding | 0 | 0 | 1
Not completed — Unknown if completed | 1 | 4 | 2
Period: In-Hospital Study Drug Infusion
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Started | 309 | 312 | 346
Completed | 214 | 229 | 266
Not Completed | 95 | 83 | 80
Not completed — Discharged | 19 | 18 | 13
Not completed — Protocol non-compliance | 14 | 17 | 10
Not completed — Withdrawal by Subject | 13 | 7 | 12
Not completed — Death or comfort care | 12 | 11 | 6
Not completed — Emergency unblinding | 11 | 4 | 7
Not completed — Seizure or concern for seizure | 8 | 9 | 17
Not completed — CVA/thrombotic event or concern for one | 5 | 5 | 4
Not completed — Required CPR | 3 | 7 | 1
Not completed — Other safety concern | 4 | 2 | 3
Not completed — Taken into police custody | 4 | 0 | 3
Not completed — Found not to be injured | 1 | 1 | 1
Not completed — Transfer to non-participating facility | 1 | 1 | 0
Not completed — Other procoagulant administered | 0 | 1 | 2
Not completed — Unknown if completed | 0 | 0 | 1
Period: 6-Month Follow-up
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Started | 309 | 312 | 346
Completed | 270 | 261 | 288
Not Completed | 39 | 51 | 58
Not completed — Withdrawal by Subject | 25 | 25 | 26
Not completed — Calls unreturned or refused contact | 4 | 15 | 20
Not completed — No contact information | 5 | 6 | 5
Not completed — Homeless | 4 | 3 | 6
Not completed — Prisoner at time of enrollment | 0 | 0 | 1
Not completed — Prisoner at time of follow-up | 0 | 2 | 0
Not completed — Patient at psychiatric hospital | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects for whom study drug administration was started minus one Bolus Only arm subject who was mistakenly enrolled while in police custody.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only | Total
Number analyzed (Participants) | 309 | 312 | 345 | 966
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [25 to 55] | 39 [26 to 57] | 40 [26 to 56] | 38 [25 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 85 | 90 | 251
  Male | 233 | 227 | 255 | 715
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was not reported at Canadian sites.
  Participants
    Hispanic or Latino | 40 | 40 | 43 | 123
    Not Hispanic or Latino | 225 | 224 | 251 | 700
    Unknown or Not Reported | 44 | 48 | 51 | 143
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was not reported at Canadian sites.
  Participants
    American Indian or Alaska Native | 2 | 4 | 4 | 10
    Asian | 7 | 13 | 10 | 30
    Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 3
    Black or African American | 46 | 50 | 53 | 149
    White | 213 | 202 | 227 | 642
    More than one race | 2 | 3 | 0 | 5
    Unknown or Not Reported | 38 | 39 | 50 | 127
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 28 | 36 | 88
  United States | 285 | 284 | 309 | 878
Penetrating injury [Count of Participants; unit: Participants] | 16 | 12 | 5 | 33
Cause of injury [Count of Participants; unit: Participants] — Population: Cause of injury missing on 1 placebo participant and 5 bolus only participants.
  Participants
    number analyzed (Participants) | 308 | 312 | 340 | 960
    Motor vehicle occupant | 113 | 103 | 115 | 331
    Motor vehicle motorcycle | 33 | 32 | 44 | 109
    Motor vehicle bicycle/pedestrian | 56 | 61 | 62 | 179
    Fall at ground level | 37 | 44 | 45 | 126
    Fall at more than 1 meter | 32 | 40 | 38 | 110
    Assault | 24 | 20 | 25 | 69
    Suicide | 9 | 8 | 5 | 22
    Other | 4 | 4 | 6 | 14
Prehospital Glasgow Coma Scale [Count of Participants; unit: Participants] — Neurological scale used to assess the level of consciousness following traumatic brain injury. Scores range from 3 to 15. Scores of 3-8 are generally considered severe, 9-12 moderate, and 13-15 minor.
  Participants
    3-8 | 186 | 169 | 177 | 532
    9-12 | 115 | 129 | 159 | 403
    13-15 | 8 | 14 | 9 | 31
Injury Severity Score (ISS) [Median (Inter-Quartile Range); unit: score on a scale] — The Injury Severity Score is a measure used to assess trauma severity. It is correlated with mortality, morbidity, and hospital length of stay. The score ranges between 0 (no injury) and 75 (unsurvivable injury). Scores greater than 15 are defined as major trauma. Population: ISS is sometimes not available if the patient dies early or there is insufficient information about injuries in specific body regions. The measure is missing for 7 placebo, 8 bolus-maintenance, and 3 bolus only participants.
  score on a scale
    number analyzed (Participants) | 302 | 304 | 342 | 948
    (all) | 17 [9 to 27] | 17 [8 to 27] | 17 [8 to 27] | 17 [9 to 27]
Head Abbreviated Injury Score (AIS) [Count of Participants; unit: Participants] — The Abbreviated Injury Scale is an anatomical-based coding system used to classify and describe the severity of injuries. The scores for a particular region range from 0 (no injury) to 6 (unsurvivable injury). Population: Head AIS is sometimes not available if the patient dies early or there is insufficient information about injuries to the head. The measure is missing for 8 placebo, 6 bolus-maintenance, and 1 bolus only participants.
  Participants
    number analyzed (Participants) | 301 | 306 | 344 | 951
    0-1 | 76 | 86 | 103 | 265
    2 | 46 | 48 | 48 | 142
    3 | 61 | 64 | 66 | 191
    4 | 67 | 56 | 71 | 194
    5-6 | 51 | 52 | 56 | 159

OUTCOME MEASURES:

1. Primary Outcome: Dichotomized Glasgow Outcome Scale Extended (GOS-E) at 6 Months
Description: GOS-E subdivides the categories of severe and moderate disability and good recovery using a scale of 1 to 8 where 1 = death, 2 = vegetative state, 3 = lower severe disability, 4 = upper severe disability, 5 = lower moderate disability, 6 = upper moderate disability, 7 = lower good recovery, and 8 = upper good recovery. Structured telephone interviews have been developed and validated for the GOS-E and these questions were incorporated into the follow-up survey. GOS-E was dichotomized into unfavorable (1 to 4) and favorable (5 to 8) outcomes.
Time Frame: 6 months post-injury
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Combined TXA Arms: Includes both the Bolus-Maintenance (1 gram IV TXA bolus in the prehospital setting followed by a 1 gram IV maintenance infusion initiated on hospital arrival and infused over 8 hours) and Bolus Only (2 grams IV TXA bolus in the prehospital setting followed by a placebo maintenance infusion initiated on hospital arrival and infused over 8 hours) treatment arms.
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only | Combined TXA Arms
Number analyzed (Participants) | 309 | 312 | 345 | 657
Participants
  Unfavorable GOS-E (<=4) | 107 | 108 | 110 | 218
  Favorable GOS-E (>4) | 163 | 153 | 178 | 331
  Missing GOS-E | 39 | 51 | 57 | 108
Statistical Analysis 1: Comparison: Placebo vs Combined TXA Arms; This study was designed with an asymmetric boundary for tests for treatment harm and benefit. The conventional 0.025 level was used to test for harm while a 0.1 level was used to determine benefit for this Phase II trial. Statistical significance for the primary analysis was conducted under a group-sequential design that included a single, interim futility analysis using a Wang-Tsiatis boundary with parameter 0.8 based on outcome data from the first 200 subjects; Test type: Superiority; p = .1809, Regression, Logistic — Based on an interim futility analysis, a one-sided P-value less than .1028 was required to declare benefit; Analysis was adjusted for regional site. Missing outcomes were multiply imputed; Odds Ratio (OR) = 0.87 — Odds ratio for unfavorable GOS-E (<=4) for the Combined TXA Arms (numerator) vs. Placebo (denominator)

2. Secondary Outcome: Number of Participants Who Died Within 28 Days
Description: The counts of patients who died on or before day 28 are reported.
Time Frame: 28 days after hospital arrival
Population: Subjects for whom study drug administration was started and 28-day vital status was definitively obtained. Patients excluded from the counts include subjects who withdrew from the study prior to day 28 and subjects who were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 285 | 285 | 318
Participants | 50 | 53 | 40

3. Secondary Outcome: Disability Rating Scale (DRS) at 6 Months
Description: The DRS is designed to classify patients based on their degree of function after brain injury. The DRS consists of 8 items that fall into 4 categories: (a) arousability, awareness and responsivity, (b) cognitive ability for self-care activities, (c) dependence on others, and (d) psychosocial adaptability. The score ranges from 0 (no disability) to 30 (death).
Time Frame: 6 months post-injury
Population: Subjects for whom study drug administration was started and DRS questions were obtained at 6 months. Excluded subjects include those who withdrew prior to 6 months after injury and those lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 266 | 261 | 287
score on a scale | 8.0 (11.8) | 8.1 (11.9) | 6.6 (10.8)

4. Secondary Outcome: Number of Participants With Unfavorable Outcome on Dichotomized Glasgow Outcome Scale Extended (GOS-E) at Discharge
Description: GOS-E subdivides the categories of severe and moderate disability and good recovery using a scale of 1 to 8 where 1 = death, 2 = vegetative state, 3 = lower severe disability, 4 = upper severe disability, 5 = lower moderate disability, 6 = upper moderate disability, 7 = lower good recovery, and 8 = upper good recovery. Structured telephone interviews have been developed and validated for the GOS-E and these questions were incorporated into the follow-up survey. GOS-E was dichotomized into unfavorable (1 to 4) and favorable (5 to 8) outcomes. The number of subjects with unfavorable outcome is reported.
Time Frame: At the end of the hospital stay (average of 9 days post injury)
Population: Subjects for whom study drug administration was started and for whom Glasgow Outcome Score Extended was obtained at discharge. Subjects who withdrew prior to discharge make up most of the subjects who were excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 292 | 294 | 329
Participants | 196 | 193 | 228

5. Secondary Outcome: Disability Rating Scale (DRS) at Discharge
Description: as for outcome 3
Time Frame: At the end of the hospital stay (average of 9 days post injury)
Population: Subjects for whom study drug administration was started and for whom discharge Disability Rating Scale was obtained. Subjects who withdrew prior to discharge make up most of the subjects who were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 291 | 294 | 329
score on a scale | 9.0 (11.1) | 9.4 (11.0) | 8.1 (9.8)

6. Secondary Outcome: Number of Participants With Intracranial Hemorrhage (ICH) Progression
Description: All clinically indicated head computed tomography (CT) scans obtained during the initial hospitalization or within the first 28 days were assessed for ICH. Parenchymal (IPH), subdural (SDH) and epidural (EDH) hemorrhage volumes were measured and quantified using volumetric software and verified by manual calculations based on the previously validated ABC/2 technique. The sum of the IPH, SDH, and EDH volumes were compared across scans. A relative increase of 33% (and at least a 1 ml increase) on any subsequent scan compared to the initial scan was defined as a progression.
Time Frame: From hospital admission through 28 days or the end of the hospital stay if sooner (average of 13 days among patients with multiple scans)
Population: Subjects for whom study drug administration was started and for whom two or more analyzable head CT scans were obtained prior to a hematoma evacuation. Excluded subjects primarily include those who died or withdrew before an initial or second CT scan was taken, who had a hematoma evacuation prior to a second scan, or who had only one negative CT.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 148 | 154 | 178
Participants | 30 | 26 | 27

7. Secondary Outcome: Marshall Computed Tomography (CT) Score on Initial Head CT
Description: The Marshall classification categorizes patients into one of six categories (I to VI) of increasing severity on the basis of findings on non-contrast CT scan of the brain. Higher categories have worse prognosis and survival.
Time Frame: Initial head CT (average of 1.9 hours post-injury)
Population: Subjects who received an initial head computed tomography scan with sufficient information to be scored.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 291 | 290 | 332
Participants
  Diffuse injury I | 120 | 115 | 134
  Diffuse injury II | 106 | 117 | 135
  Diffuse injury III | 12 | 12 | 12
  Diffuse injury IV | 7 | 4 | 5
  Mass lesion V/VI | 46 | 42 | 46

8. Secondary Outcome: Rotterdam Computed Tomography (CT) Score Among Subjects With Intracranial Hemorrhage (ICH) on Initial Head CT
Description: The Rotterdam classification includes four independently scored elements: degree of basal cistern compression, degree of midline shift, presence of epidural hematomas, and presence of intraventricular or subarachnoid blood. The elements are combined to form an overall score from 1 to 6 with higher scores having worse prognosis and survival.
Time Frame: Initial head CT (average of 1.9 hours post-injury)
Population: Subjects determined by the central image reviewer to have an intracranial hemorrhage (ICH) on the initial head computed tomography (CT) scan and sufficient information to assign the Rotterdam score.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 158 | 161 | 187
Participants
  1 | 2 | 1 | 5
  2 | 32 | 28 | 36
  3 | 81 | 91 | 98
  4 | 17 | 24 | 28
  5 | 21 | 12 | 17
  6 | 5 | 5 | 3

9. Secondary Outcome: Number of Participants With One or More Neurosurgical Interventions
Description: Neurosurgical interventions include craniotomy, craniectomy, and placement of a neuromonitoring or drainage device. Counts are of subjects with one or more neurosurgical interventions.
Time Frame: From hospital admission through 28 days or the end of the hospital stay if sooner (average of 9 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 309 | 312 | 345
Participants | 54 | 62 | 75

10. Secondary Outcome: Hospital-free Days
Description: Hospital-free days count any day from hospital admission through day 28 that the patient is alive and out of the hospital.
Time Frame: From hospital admission through day 28
Population: Subjects for whom study drug administration was started and for whom discharge status was known. Subjects who withdrew prior to discharge make up most of the subjects who were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 295 | 292 | 331
days | 13.6 (10.7) | 13.6 (10.7) | 14.1 (10.4)

11. Secondary Outcome: Intensive Care Unit (ICU)-Free Days
Description: ICU-free days count any day from hospital admission through day 28 that the patient is alive and not in the ICU. Subjects who die prior to discharge (even if after 28 days) are assigned a value of 0.
Time Frame: From hospital admission through day 28
Population: Subjects for whom study drug administration was started and for whom number of ICU days through 28 days was known. Subjects who withdrew prior to discharge make up most of the subjects who were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 295 | 293 | 331
days | 18.5 (10.6) | 18.1 (10.8) | 19.1 (9.7)

12. Secondary Outcome: Ventilator-free Days
Description: Ventilator-free days count any day from hospital admission through day 28 that the patient is alive and does not require mechanical ventilatory support. Subjects who die prior to discharge (even if after 28 days) are assigned a value of 0.
Time Frame: From hospital admission through day 28
Population: Subjects for whom study drug administration was started and for whom number of ventilator days through 28 days was known. Subjects who withdrew prior to discharge make up most of the subjects who were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 295 | 293 | 331
days | 20.2 (10.5) | 19.9 (10.8) | 20.9 (9.7)

13. Secondary Outcome: Number of Participants With Seizure
Description: Seizures may cause involuntary changes in body movement or function, sensation, awareness, or behavior. Seizures are often associated with a sudden and involuntary contraction of a group of muscles and loss of consciousness. Seizures or episodes of seizure-like activity were reported by medics in the field following the start of study drug infusion through hand-off to the trauma center and by trauma center staff through discharge. Reported events were included if providers gave anti-seizure medication and/or the event was confirmed by EEG.
Time Frame: From start of study drug infusion through 28 days or the end of the hospital stay if sooner (average of 9 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 309 | 312 | 345
Participants | 7 | 5 | 17

14. Secondary Outcome: Number of Participants With Cerebral Ischemic Event
Description: Diagnosis of cerebral ischemic event
Time Frame: From hospital admission through 28 days or the end of the hospital stay if sooner (average of 9 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 309 | 312 | 345
Participants | 10 | 3 | 13

15. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: Diagnosis of an acute myocardial infarction
Time Frame: From hospital admission through 28 days or the end of the hospital stay if sooner (average of 9 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 309 | 312 | 345
Participants | 1 | 3 | 2

16. Secondary Outcome: Number of Participants With Deep Vein Thrombosis (DVT)
Description: Diagnosis of DVT
Time Frame: From hospital admission through 28 days or the end of the hospital stay if sooner (average of 9 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 309 | 312 | 345
Participants | 9 | 3 | 10

17. Secondary Outcome: Number of Participants With Pulmonary Embolus (PE)
Description: Diagnosis of PE
Time Frame: From hospital admission through 28 days or the end of the hospital stay if sooner (average of 9 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 309 | 312 | 345
Participants | 5 | 3 | 6

18. Secondary Outcome: Number of Participants With Any Thromboembolic Event
Description: Diagnosis of one or more of the following: cerebral ischemic event, myocardial infarction (MI), deep vein thrombosis (DVT), pulmonary embolism (PE), or any other thromboembolic event
Time Frame: From hospital admission through 28 days or the end of the hospital stay if sooner (average of 9 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 309 | 312 | 345
Participants | 30 | 13 | 31

19. Other Pre Specified Outcome: Fibrinolysis at Hospital Admission
Description: Alterations in fibrinolysis based on fibrinolytic pathway mediators and degree of clot lysis based on kaolin-activated thromboelastography (TEG) and defined as LY30 or the per cent lysis that occurs 30 minutes after maximum amplitude (MA) is achieved. LY30 is categorized as <0.8% (fibrinolysis shutdown), 0.8-3% (normal), and >3% (hyperfibrinolysis).
Time Frame: First blood draw (average of 1.6 hours post-injury)
Population: Subjects with an LY30 measurement at hospital admission are included. Subjects who were transported to trauma centers without a TEG machine, who died prior to the initial blood draw, or who withdrew or refused a blood draw were excluded. Additional exclusions included blood draw missed by study staff and technical difficulties with processing.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
Number analyzed (Participants) | 240 | 246 | 261
Participants
  <0.8 (fibrinolysis shutdown) | 148 | 157 | 165
  0.8-3% (normal) | 56 | 61 | 65
  >3% (hyperfibrinolysis) | 36 | 28 | 31

ADVERSE EVENTS:
Time Frame: Adverse events data were captured from the beginning of study drug infusion on day 0 through day 28. While follow-up time varies by patient due to withdrawals, transfers to non-participating hospitals, deaths, and participants lost to follow-up, all analysis patients were "at risk" for adverse events during at least some period of time and are thus included in all adverse event denominators.
Description: Chart reviews were made daily. Events prespecified as possibly related to study drug were categorized for seriousness by site PIs and are listed in both the "Serious" and "Other" AE sections below. Other events (marked with "^") were monitored and reported but not considered adverse events of the study drug. These are listed in the "Other" AE section since they were not assessed for seriousness. One Bolus Only arm subject who was mistakenly enrolled while in police custody is excluded.
Arm/Group | Placebo | Bolus-Maintenance | Bolus Only
All-Cause Mortality (participants affected / at risk) | 50/309 | 53/312 | 40/345
Serious Adverse Events (participants affected / at risk) | 25/309 | 13/312 | 24/345
Other Adverse Events (participants affected / at risk) | 81/309 | 74/312 | 92/345
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=309) | Bolus-Maintenance (N=312) | Bolus Only (N=345)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (MI) (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Cerebrovascular accident - hemorrhagic (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Cerebrovascular accident - thrombotic (Nervous system disorders) | 9 (10) | 1 (1) | 11 (11)
Seizures (Nervous system disorders) | 2 (2) | 3 (3) | 6 (6)
Pulmonary embolism (PE) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 4 (4)
Cerebral vascular emboli (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebral venus sinus thrombosis (Vascular disorders) | 4 (4) | 0 (0) | 4 (4)
Deep vein thrombosis (DVT) (Vascular disorders) | 4 (5) | 1 (1) | 5 (5)
Embolic infarcts (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Inferior vena cava thrombus (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Internal jugular vein thrombus (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular thrombus (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=309) | Bolus-Maintenance (N=312) | Bolus Only (N=345)
Cardiac arrest (non-fatal)^ (Cardiac disorders) | 5 (5) | 5 (5) | 2 (2)
Cardiac failure^ (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (MI) (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Pseudomembranous colitis^ (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
Abdominal Compartment Syndrome^ (General disorders) | 0 (0) | 1 (1) | 0 (0)
Central diabetes insipidus^ (General disorders) | 5 (5) | 0 (0) | 4 (4)
Cerebral vasospams^ (General disorders) | 4 (4) | 2 (2) | 4 (4)
Extremity Compartment Syndrome^ (General disorders) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis^ (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Liver failure^ (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bloodstream infection^ (Infections and infestations) | 1 (1) | 4 (4) | 3 (3)
Empyema^ (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Intra-abdominal abscess^ (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Meningitis^ (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia^ (Infections and infestations) | 29 (29) | 36 (36) | 45 (45)
Sepsis^ (Infections and infestations) | 6 (6) | 11 (11) | 9 (9)
Urinary tract infection (UTI)^ (Infections and infestations) | 9 (9) | 15 (15) | 9 (9)
Wound infection^ (Infections and infestations) | 3 (3) | 0 (0) | 5 (5)
Hypernatremia^ (Metabolism and nutrition disorders) | 10 (10) | 8 (8) | 14 (14)
Cerebrovascular accident - hemorrhagic (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Cerebrovascular accident - thrombotic (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2)
Seizures (Nervous system disorders) | 5 (5) | 2 (2) | 11 (11)
Acute kidney injury (AKI)^ (Renal and urinary disorders) | 13 (13) | 17 (17) | 16 (16)
Renal failure^ (Renal and urinary disorders) | 0 (0) | 0 (0) | 5 (5)
Acute Respiratory Distress Syndrome (ARDS)^ (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 8 (8) | 5 (5)
Pulmonary embolism (PE) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Cerebral venus sinus thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 3 (3)
Deep vein throbosis (DVT) (Vascular disorders) | 5 (5) | 2 (2) | 5 (5)
Superficial venus thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Protocol in force at beginning of enrollment (2015-04-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT01990768/Prot_SAP_ICF_000.pdf
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Protocol after Amendment 2 (2015-07-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT01990768/Prot_SAP_ICF_001.pdf
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Protocol after Amendment 2.1 (2016-08-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT01990768/Prot_SAP_ICF_002.pdf